CLINICAL TRIAL: NCT05705817
Title: Assistive Soft Skills and Employment Training (ASSET) in Traumatic Brain Injury
Brief Title: Assistive Soft Skills and Employment Training (ASSET) in TBI Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-1201-22
Record Dates: First submitted 2023-01-09; First posted 2023-01-31 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Behavioral: Assistive Soft Skills and Employment Training (ASSET)

INTERVENTIONS:
Behavioral: Assistive Soft Skills and Employment Training (ASSET) — The ASSET program is a 15-session training program that combines specific skill training, structured learning, social performance training and a social hour to practice skills through a manualized group intervention. Specific skills taught within the program include communication, enthusiasm and attitude, teamwork, networking, problem-solving and critical thinking, and professionalism.

SUMMARY:
Pediatric traumatic brain injury (TBI) is often associated with difficulties in social functioning. Loss of social contacts and difficulties maintaining social connections is common after pediatric TBI, extending into adulthood. Social skills are a key aspect of social functioning critical to forming and maintaining social relationships with others, including family, friends, teachers and co-workers. Social skills deficits are thus critical to social participation and overall quality of life. The identification of treatment techniques to effectively address these issues are thus of paramount importance. The ability to improve social skills in adolescents and young adults is critical as they transition from school settings into the workforce. Impairments in social skills have been demonstrated to underlie difficulties transitioning from school to work and independent living in students with disabilities. Therefore, targeting social skills interventions as individuals enter adulthood and enter the workforce is likely to improve overall functioning during this transitional period in their lives.

The current study will examine preliminary efficacy of a manualized group intervention that targets social skills, specifically work-related social skills known as soft skills. Targeting not only general social skills, but soft skills in particular, is expected to be particularly useful for teens and young adults as they transition from school into the workforce.

The Assistive Soft Skills and Employment Training (ASSET) is a 15-session training program that combines specific skill training, structured learning, social performance training and a social hour to practice skills through a manualized group intervention. Specific skills taught within the program include communication, attitude and enthusiasm, teamwork, networking, problem-solving and critical thinking, professionalism, mental health and stress management, awareness of self and others, workplace relationships and self-advocacy. ASSET utilizes a manualized curriculum and provides additional support including handouts, PowerPoint summaries, instructional procedures, video models, materials for caregivers, and an online platform to support learning the program. ASSET has been utilized with young adults with ASD with very positive results, improving performance on measures of social skills, social communication, self-confidence/self-efficacy and psychological wellness. The current proposal will test the efficacy of the ASSET program in youth and young adults with TBI between the ages of 15 and 25, a critical time as individuals' transition from school settings into the workforce. The proposal will evaluate the primary outcome of improvements in social skills following completion of the ASSET program. Secondary outcomes of self-efficacy, depression, anxiety and quality of life will also be evaluated following completion of the program.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-25
* At least one year post injury.

Exclusion Criteria:

* any other significant neurological history other than their TBI.
* unstable or uncontrolled seizures (as defined by an increase in the rate of seizures over the 3 months before study participation)

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Social Skills Questionnaire for Traumatic Brain Injury | Within 2 weeks
  This is a 41-tem scale to assess social skills in TBI

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Lengenfelder, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No